CLINICAL TRIAL: NCT03605225
Title: Development and Validation of an Android-based Application for Anaesthesia Neuromuscular Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: APP NMM
Record Dates: First submitted 2018-07-20; First posted 2018-07-30 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Neuromuscular Blockade; Neuromuscular Monitoring
Keywords: Android application; Anesthesia; intraoperative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cellphone application (Experimental): Train of Four (TOF) ratio displayed by the Cellphone Application
  Interventions: Device: mobile cellphone application test
- Draeger TOF Scan (Active Comparator): Train of Four (TOF) ratio displayed by the Draeger TOF Scan
  Interventions: Device: mobile cellphone application test

INTERVENTIONS:
Device: mobile cellphone application test — Placement of cellphone on the patient´s hand and recording accelerometric data during elicited muscular contractions.

SUMMARY:
The present study aims to assess the accuracy of a newly developed Android Smartphone Application in measuring the degree of Neuromuscular block in the perioperative period.

This will be achieved by comparing Train-of-four Ratio measurements using this application with those obtained from a standard commercialized neuromuscular monitor.

DETAILED DESCRIPTION:
Since Harold Randall Griffith pioneered by the use of curare during anaesthesia by administering it to a young man during an appendectomy in Montreal, the practice of anaesthesiology has completely changed and the world of Neuromuscular Blocking has been thoroughly fine-tuned: increased knowledge and clinical experience, development of new Neuromuscular Blocking Agents (NMBA) with fewer side-effects and well-studied pharmacokinetic profiles, introduction of new antagonizing drugs such as Sugammadex, as well as refinement of neuromuscular block measuring instruments. NMBAs are routinely administered to patients in a multiplicity of anaesthetic settings, and the possibility and availability of instruments allowing the accurate measurement of the degree of neuromuscular block has raised the standards of their use and reversal. The absence of a residual neuromuscular blockade is now widely considered an anesthetic must, as incomplete recovery has been long-established as a strong contributor to post-anesthesia morbidity and mortality. Considering the proven inconsistent, inter/intra-variable and inaccurate character of the human senses to estimate adequate neuromuscular recovery after NMBA use, the proper assessment of neuromuscular recovery can only be done by means of objective methods.3 For this purpose, one of the most widely used methods is the Train of Four (TOF): transcutaneous application of a series of 4 square-wave supra-maximal electrical stimuli over the course of a nerve of choice (most commonly the ulnar nerve). These are applied at a frequency of 2Hz, and each with a duration of 0,2ms. These stimuli elicit a motor response on the adductor pollicis muscle, which on its turn dictates the abduction of the thumb. The acceleration of this movement can be followed by means of an uni/multi-directional accelerometer attached to the thumb. The ratio of the acceleration of the 4th and 1st elicited contractions is called the TOF-Ratio, and this TOF-ratio is a clinically and scientifically established method of assessing neuromuscular block recovery. A value of 1 translates a full recovery of the muscular function of a patient. In modern Anesthesia, the bar for deeming a recovery as adequate has been set at a minimum of a TOF-Ratio of >0.9, with some authors advocating a ratio of 1 as the only acceptable and complications-avoiding result.

Although an effective measurement of muscular recovery parameters is necessary, daily clinical limitations dictate other practices. Medical devices are expensive and not always available for immediate use. Some devices are also only able to deliver the electrical impulses, but not to measure acceleromyographic parameters. These limitations often force anaesthesiologists to undertake on-the-spot guess-practices (assuming recovery based on a particular NMBA's half-life and its last administered dose), or "d'office" actions (standard NMBA reversal) to determine if a patient has adequately recovered. These methods are inherently associated with major pitfalls/iatrogenic side-effects and are major determinants of a high post-operative morbidity and mortality.

In this study the investigators aim to assess the capability of a dedicated smartphone application to transform and incorporate a Smartphone's accelerometric data to accurately measure the TOF-Ratio in an anaesthesia setting and to compare it to commercially used and established neuromuscular block measuring devices.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiology (ASA) physical status classification I to III
* elective procedures under general anesthesia requiring use of a non-depolarizing neuromuscular blocking agent

Exclusion Criteria:

* Known or suspected central or peripheral neuropathies of any ethology
* Muscular dystrophies
* Skin burns and trauma at measurement sites (arms).
* Musculo-tendinopathies of the arms and hands.
* All conditions that might be judged to alter appropriate peripheral neuromuscular conduction.
* Fragile skin impeding placement of electrocardiogram electrodes at measurement sites.
* Allergy to ECG Electrodes
* Intra-operative position impeding proper use of any of the two used neuromuscular monitors.
* Calibration/device failure
* Failure to properly stabilize the patient's hand in supination (so that the smartphone won't dislocate itself during measurements)
* Patient premedication judged to interfere with proper cognitive assimilation of the study concept.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-11-16 (Actual)

PRIMARY OUTCOMES:
Train of Four ratio | before neuromuscular blocking drug administration, approximately 15 minutes after administration, and before extubation.
  Ratio between de fourth and first accelerometric twitches of the thumb after elicited contraction via transcutaneous electrical stimulation of the ulnar nerve.

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Carvalho, MSc, MD, Principal Investigator — Universitair Ziekenhuis Brussel; Jan D'Haese, MD, Study Chair — Universitair Ziekenhuis Brussel; Jan Poelaert, PhD, MD, Study Director — Universitair Ziekenhuis Brussel
Locations (1):
- universitair Ziekenhuis brussel, Jette, België, Belgium

REFERENCES:
- [Derived] Verdonck M, Carvalho H, Berghmans J, Forget P, Poelaert J. Exploratory Outlier Detection for Acceleromyographic Neuromuscular Monitoring: Machine Learning Approach. J Med Internet Res. 2021 May 31;23(6):e25913. doi: 10.2196/25913. PMID 34152273